CLINICAL TRIAL: NCT02642055
Title: Efficacy of NEURO+ Attention Training: A Randomized, Controlled, Blinded, Clinical Trial
Brief Title: Efficacy of Neuro+ Attention Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuro+ (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NEURO+001
Record Dates: First submitted 2015-12-18; First posted 2015-12-30 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-05

CONDITIONS: ADHD
Keywords: ADHD; Neurofeedback; Biofeedback; Neuro+; Go/no-go; Attention training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neuro+ Intervention (Experimental): 30 sessions (900 minutes) of Neuro+ Attention Training administered over 10 weeks.
  Interventions: Behavioral: Neuro+ Attention Training
- Treatment as Usual (Active Comparator): Continuation of current treatment for ADHD
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Neuro+ Attention Training — Attention training program with Neuro+ software
  Arms: Neuro+ Intervention
Other: Treatment as Usual — Continuation of current ADHD treatment
  Arms: Treatment as Usual

SUMMARY:
This study evaluates the efficacy of the Neuro+ Attention Training System (Neuro+) in improving attention skills in children. Half of participants will receive the Neuro+ intervention for 10 weeks, while the other half will continue treatment as usual (TAU) for the same period. We expect those receiving the Neuro+ intervention to see significant improvements in ADHD symptoms relative to the TAU controls.

DETAILED DESCRIPTION:
Neuro+ a non-pharmacological intervention that targets the underlying neural signatures and cognitive deficits which are assumed to mediate attention pathways. Targeting those underlying areas could reduce ADHD symptoms and potentially lead to greater transfer and generalization to functioning in the classroom and every day life.

Neuro+ combines neurofeedback, biofeedback, and go/no-go training protocols embedded in a training video game to help develop and improve attention skills. The protocols function as follows:

Neurofeedback: Users wear a dry, wireless, easy-to-use EEG headset that interfaces with computer software to provide feedback on their level of brain activation, or focus. Users must focus in order to advance through the training game.

Motion-biofeedback: Accelerometers in the headset send data on users' movement to the training game, such that users must maintain complete control of their bodies and remain absolutely still in order to advance through the game and avoid costly point penalties.

Go/no-go training: To practice impulse control, users will be challenged with adaptive "go/no-go tasks," requiring them to quickly and accurately respond to target stimuli and ignore distractions, with the tasks becoming more difficult as the user improves.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 to 13 at the time of parental informed consent.
* Confirmed ADHD diagnosis at clinic
* No usage of ADHD drugs in past 30 days, or stable on current drug regimen for at least 30 days. Drugs include: Pre specified, oral psychostimulants, including ADDERALL XR® [mixed salts of a single-entity amphetamine product], VYVANSE® [lisdexamfetamine dimesylate], CONCERTA® [methylphenidate HCl], FOCALIN XR® [dexmethylphenidate HCl], RITALIN LA® [methylphenidate HCl extended-release], METADATE CD® [methylphenidate HCl, USP], or other FDA-approved equivalents.
* Ability to follow written and verbal instructions (English)
* Girls or Boys
* Functioning at an age-appropriate level intellectually.
* Ability to comply with all the testing and requirements.

Exclusion Criteria:

* Current, controlled (requiring a restricted medication) or uncontrolled, comorbid psychiatric diagnosis with significant symptoms such as post-traumatic stress disorder, psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder, conduct disorder, or other symptomatic manifestations that in the opinion of the Investigator that may confound study data/assessments.
* Motor condition that prevents game playing.
* Recent history (within the past 6 months) of suspected substance abuse or dependence.
* History of seizures (exclusive of febrile seizures), a tic disorder, significant tics, or a current diagnosis of Tourette's Disorder.
* Taken part in a clinical trial within 30 days prior to screening.
* Diagnosis of color blindness.
* Regular use of psychoactive drugs that in the opinion of the Investigator may confound study data/assessments.
* Any other medical condition that in the opinion of the Investigator may confound study data/assessments.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in ADHD symptoms with Quotient ADHD System assessment | At screening and at final clinical visit within 1 week following intervention
  Assessments to be conducted with the Quotient ADHD System
Change in assessment of ADHD symptoms with Conners 3-Parent rating scale | At screening and at final clinical visit within 1 week following intervention
  Assessments to be conducted with the Conners 3-Parent rating scale
Incidence of adverse events | As reported by subjects at final clinical visit, which occurs within 1 week following intervention.
  Self-reported incidence of adverse events

SECONDARY OUTCOMES:
Self-reported convenience ratings of Neuro+ intervention | At final clinical visit, within 1 week following intervention
  As evaluated on a Likert scale, the extent to which subjects and parents found the Neuro+ intervention convenient/easy-to-use

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Vaishnavi, MD, PhD, Principal Investigator — Carolina Partners in Mental HealthCare, PLLC
Locations (1):
- Neuropsychiatric Clinic at Carolina Partners in Mental HealthCare, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No